CLINICAL TRIAL: NCT04153149
Title: HELIOS-B: A Phase 3, Randomized, Double-blind, Placebo-controlled, Multicenter Study to Evaluate the Efficacy and Safety of Vutrisiran in Patients With Transthyretin Amyloidosis With Cardiomyopathy (ATTR Amyloidosis With Cardiomyopathy)
Brief Title: HELIOS-B: A Study to Evaluate Vutrisiran in Patients With Transthyretin Amyloidosis With Cardiomyopathy
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Alnylam Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALN-TTRSC02-003; 2023-508366-15-00 (EU CTIS Number)
Record Dates: First submitted 2019-11-04; First posted 2019-11-06 (Actual); Results first posted 2025-10-21 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Transthyretin Amyloidosis (ATTR) With Cardiomyopathy
Keywords: ATTR; Cardiomyopathy; Amyloidosis; TTR; Transthyretin; TTR-mediated amyloidosis; Amyloidosis, Hereditary; Amyloidosis, Hereditary, Transthyretin-Related; Familial Amyloidosis; RNAi therapeutic; Transthyretin amyloid cardiomyopathy; TTR cardiomyopathy; ATTR-CM; Wild-type TTR; V122I; TTR amyloidosis; Amyloidosis, Wild Type
MeSH Terms: conditions — Amyloidosis, Hereditary, Transthyretin-Related; Cardiomyopathies; Amyloidosis; Amyloidosis, Familial

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Vutrisiran 25 mg (Experimental): Participants received vutrisiran 25 milligrams (mg) administered subcutaneously (SC) once every 3 months (q3M) during the 36-month double-blind (DB) period. After the DB period, participants continue receiving vutrisiran, 25 mg, SC injection, q3M for up to 24 months in the open-label treatment extension (OLE) period.
  Interventions: Drug: Vutrisiran
- Placebo (Placebo Comparator): Participants received vutrisiran matching placebo administered SC q3M during the 36-month DB period. After the DB period, participants receive vutrisiran, 25 mg, SC injection, q3M for up to 24 months in the OLE period.
  Interventions: Drug: Vutrisiran; Drug: Sterile Normal Saline (0.9% NaCl)

INTERVENTIONS:
Drug: Vutrisiran — Vutrisiran will be administered by SC injection.
  Other Names: ALN-TTRSC02
Drug: Sterile Normal Saline (0.9% NaCl) — Sterile normal saline (0.9% NaCl) will be administered by SC injection.
  Arms: Placebo

SUMMARY:
This study will evaluate the efficacy and safety of vutrisiran 25 mg administered subcutaneously (SC) once every 3 months (q3M) compared to placebo in participants with ATTR amyloidosis with cardiomyopathy.

ELIGIBILITY:
Inclusion Criteria:

* Has a documented diagnosis of transthyretin (ATTR) amyloidosis with cardiomyopathy, classified as either hereditary ATTR (hATTR) amyloidosis with cardiomyopathy or wild-type ATTR (wtATTR) amyloidosis with cardiomyopathy meeting pre-specified diagnostic criteria
* Has medical history of heart failure (HF) with at least 1 prior hospitalization for HF OR clinical evidence of HF

Exclusion Criteria:

* Has known primary amyloidosis or leptomeningeal amyloidosis
* Has New York Heart Association (NYHA) Class IV heart failure
* Has NYHA Class III heart failure AND is at high risk based on pre-specified criteria
* Has a polyneuropathy disability (PND) Score IIIa, IIIb, or IV at the Screening visit
* Has estimated glomerular filtration rate (eGFR) <30 mL/min/1.73 m^2
* Has received prior TTR-lowering treatment
* Has other non-TTR cardiomyopathy, hypertensive cardiomyopathy, cardiomyopathy due to valvular heart disease, or cardiomyopathy due to ischemic heart disease

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 655 (Actual)
Dates: Start 2019-11-26 (Actual); Primary Completion 2024-05-08 (Actual); Study Completion 2026-12-02 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Alnylam Pharmaceuticals
Locations (109):
- United States (16):
  - Clinical Trial Site, La Mesa, California
  - Clinical Trial Site, Los Angeles, California
  - Clinical Trial Site, Stanford, California
  - Clinical Trial Site, Washington D.C., District of Columbia
  - Clinical Trial Site, Gainesville, Georgia
  - Clinical Trial Site, Chicago, Illinois
  - Clinical Trial Site, Evanston, Illinois
  - Clinical Trial Site, Boston, Massachusetts
  - Clinical Trial Site, Rochester, Minnesota
  - Clinical Trial Site, Manhasset, New York
  - Clinical Trial Site, New York, New York
  - Clinical Trial Site, Durham, North Carolina
  - Clinical Trial Site, Cleveland, Ohio
  - Clinical Trial Site, Allentown, Pennsylvania
  - Clinical Trial Site, Philadelphia, Pennsylvania
  - Clinical Trial Site, Houston, Texas
- Argentina (3):
  - Clinical Trial Site, Buenos Aires, Ciudad Autónoma de BuenosAires
  - Clinical Trial Site, Buenos Aires, Pilar
  - Clinical Trial Site, Buenos Aires
- Australia (5):
  - Clinical Trial Site, Darlinghurst, New South Wales
  - Clinical Trial Site, Northmead, New South Wales
  - Clinical Trial Site, Woolloongabba, Queensland
  - Clinical Trial Site, Adelaide, South Australia
  - Clinical Trial Site, Melbourne, Victoria
- Austria (2):
  - Clinical Trial Site, Graz
  - Clinical Trial Site, Vienna
- Belgium (4):
  - Clinical Trial Site, Dendermonde, Oost-Vlaanderen
  - Clinical Trial Site, Ghent, Oost-Vlaanderen
  - Clinical Trial Site, Brussels
  - Clinical Trial Site, Leuven
- Canada (2):
  - Clinical Trial Site, Toronto, Ontario
  - Clinical Trial Site, Québec, Quebec
- Clinical Trial Site, Zagreb, Croatia
- Czechia (2):
  - Clinical Trial Site, Olomouc, Olomoucký kraj
  - Clinical Trial Site, Prague, Praha, Hlavní Mesto
- Denmark (2):
  - Clinical Trial Site, Odense, Region Syddanmark
  - Clinical Trial Site, Aarhus N
- France (4):
  - Clinical Trial Site, Créteil
  - Clinical Trial Site, Marseille
  - Clinical Trial Site, Paris
  - Clinical Trial Site, Toulouse
- Germany (7):
  - Clinical Trial Site, Frankfurt am Main, Hesse
  - Clinical Trial Site, Leipzig, Saxony
  - Clinical Trial Site, Essen
  - Clinical Trial Site, Göttingen
  - Clinical Trial Site, Heidelberg
  - Clinical Trial Site, Münster
  - Clinical Trial Site, Würzburg
- Hungary (2):
  - Clinical Trial Site, Budapest
  - Clinical Trial Site, Szeged
- Clinical Trial Site, Dublin, Ireland
- Israel (3):
  - Clinical Trial Site, Haifa
  - Clinical Trial Site, Jerusalem
  - Clinical Trial Site, Ramat Gan
- Japan (12):
  - Clinical Trial Site, Tsurumai-cho, Aichi-ken
  - Clinical Trial Site, Fukuoka, Fukuoka
  - Clinical Trial Site, Kurume, Fukuoka
  - Clinical Trial Site, Kita-gun, Kagawa-ken
  - Clinical Trial Site, Nankoku, Kochi
  - Clinical Trial Site, Matsumoto, Nagano
  - Clinical Trial Site, Kashihara, Nara
  - Clinical Trial Site, Suita, Osaka
  - Clinical Trial Site, Bunkyo-ku, Tokyo
  - Clinical Trial Site, Shinjuku-Ku, Tokyo
  - Clinical Trial Site, Fukuoka
  - Clinical Trial Site, Kumamoto
- Clinical Trial Site, Riga, Latvia
- Clinical Trial Site, Hamra, Beyrouth, Lebanon
- Clinical Trial Site, Kaunas, Lithuania
- Malaysia (2):
  - Clinical Trial Site, Kuantan, Pahang
  - Clinical Trial Site, Sungai Buloh, Selangor
- Clinical Trial Site, Chisinau, Moldova
- Netherlands (3):
  - Clinical Trial Site, Eindhoven
  - Clinical Trial Site, Groningen
  - Clinical Trial Site, Utrecht
- Clinical Trial Site, Oslo, Norway
- Peru (2):
  - Clinical Trial Site, San Isidro, Lima region
  - Clinical Trial Site, Lima
- Poland (5):
  - Clinical Trial Site, Wroclaw, Lower Silesian Voivodeship
  - Clinical Trial Site, Lodz, Lódzkie
  - Clinical Trial Site, Warsaw, Masovian Voivodeship
  - Clinical Trial Site, Gdansk, Pomeranian Voivodeship
  - Clinical Trial Site, Katowice
- Portugal (5):
  - Clinical Trial Site, Lisbon, Lisbon District
  - Clinical Trial Site, Coimbra
  - Clinical Trial Site, Faro
  - Clinical Trial Site, Guimarães
  - Clinical Trial Site, Porto
- Saudi Arabia (2):
  - Clinical Trial Site, Mecca, Mecca Region
  - Clinical Trial Site, Riyadh
- Clinical Trial Site, Ljubljana, Slovenia
- Clinical Trial Site, Seoul, South Korea
- Spain (6):
  - Clinical Trial Site, L'Hospitalet de Llobregat, Barcelona
  - Clinical Trial Site, Majadahonda, Madrid
  - Clinical Trial Site, Barcelona
  - Clinical Trial Site, Bilbao
  - Clinical Trial Site, Huelva
  - Clinical Trial Site, Málaga
- Sweden (2):
  - Clinical Trial Site, Göteborg, Västerbotten County
  - Clinical Trial Site, Gothenburg
- Clinical Trial Site, Chiang Mai, Thailand
- United Kingdom (8):
  - Clinical Trial Site, Bellshill, Lanarkshire
  - Clinical Trial Site, London, London, City of
  - Clinical Trial Site, Londonderry, Londonderry
  - Clinical Trial Site, Hexham, Northumberland
  - Clinical Trial Site, Birmingham
  - Clinical Trial Site, Cardiff
  - Clinical Trial Site, London
  - Clinical Trial Site, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Access to Anonymized individual participant data that support these results is made available 12 months after study completion and not less than 12 months after the product and indication have been approved in the US and/or the EU.
  Access to data may be declined where there is likelihood a patient could be identified or other feasibility issue, where there is a potential conflict of interest, a planned business activities or an actual or potential competitive risk. Data will be provided contingent upon the approval of a research proposal and the execution of a data sharing agreement. Timeframes for data access may vary and can take up to 6 months or more.
  Requests for access to data can be submitted via the website www.vivli.org. Questions can also be directed to datasharing@alnylam.com.

REFERENCES:
- [Derived] Claggett BL, Fontana M, Vaduganathan M, Hamatani Y, Maurer MS, Gillmore JD, Solomon SD. Timing of Mortality Benefit in Outcomes Trials in Transthyretin Amyloidosis. J Am Coll Cardiol. 2025 Sep 25:S0735-1097(25)09374-X. doi: 10.1016/j.jacc.2025.09.1512. Online ahead of print. PMID 41225306
- [Derived] Jering KS, Fontana M, Lairez O, Longhi S, Azevedo O, Morbach C, Bender S, Jay PY, Vest J, Bulwer BE, Prasad N, Solomon SD, Skali H. Effects of vutrisiran on cardiac structure and function in patients with transthyretin amyloidosis with cardiomyopathy: secondary outcomes of the HELIOS-B trial. Nat Med. 2025 Oct;31(10):3560-3568. doi: 10.1038/s41591-025-03851-z. Epub 2025 Aug 6. PMID 40770082
- [Derived] Maurer MS, Berk JL, Damy T, Sheikh FH, Gonzalez-Costello J, Morbach C, Delgado D, Bondue A, Azevedo O, Poulsen SH, Jankowska EA, Yang L, Bender S, Eraly SA, Jay PY, Vest J, Fontana M. Impact of Vutrisiran on Cardiac Biomarkers in Patients With Transthyretin Amyloidosis With Cardiomyopathy From HELIOS-B. J Am Coll Cardiol. 2025 Aug 12;86(6):459-475. doi: 10.1016/j.jacc.2025.04.055. PMID 40769675
- [Derived] Witteles RM, Garcia-Pavia P, Damy T, Grogan M, Sheikh FH, Morbach C, Bender S, Exter J, Eraly SA, Fontana M. Vutrisiran Improves Survival and Reduces Cardiovascular Events in ATTR Amyloid Cardiomyopathy: HELIOS-B. J Am Coll Cardiol. 2025 Apr 30:S0735-1097(25)06170-4. doi: 10.1016/j.jacc.2025.04.008. Online ahead of print. PMID 40380962
- [Derived] Maurer MS, Witteles RM, Garcia-Pavia P, Sheikh FH, Morbach C, Rodriguez Duque D, Aldinc E, Eraly SA, Gillmore JD. Impact of Heart Failure Severity on Vutrisiran Efficacy in Transthyretin Amyloidosis With Cardiomyopathy. J Am Coll Cardiol. 2025 May 27;85(20):1927-1939. doi: 10.1016/j.jacc.2025.03.477. Epub 2025 Mar 17. PMID 40099776
- [Derived] Fontana M, Maurer MS, Gillmore JD, Bender S, Aldinc E, Eraly SA, Jay PY, Solomon SD. Outpatient Worsening Heart Failure in Patients With Transthyretin Amyloidosis With Cardiomyopathy in the HELIOS-B Trial. J Am Coll Cardiol. 2025 Feb 25;85(7):753-761. doi: 10.1016/j.jacc.2024.11.015. Epub 2024 Nov 18. PMID 39566871
- [Derived] Fontana M, Berk JL, Gillmore JD, Witteles RM, Grogan M, Drachman B, Damy T, Garcia-Pavia P, Taubel J, Solomon SD, Sheikh FH, Tahara N, Gonzalez-Costello J, Tsujita K, Morbach C, Pozsonyi Z, Petrie MC, Delgado D, Van der Meer P, Jabbour A, Bondue A, Kim D, Azevedo O, Hvitfeldt Poulsen S, Yilmaz A, Jankowska EA, Algalarrondo V, Slugg A, Garg PP, Boyle KL, Yureneva E, Silliman N, Yang L, Chen J, Eraly SA, Vest J, Maurer MS; HELIOS-B Trial Investigators. Vutrisiran in Patients with Transthyretin Amyloidosis with Cardiomyopathy. N Engl J Med. 2025 Jan 2;392(1):33-44. doi: 10.1056/NEJMoa2409134. Epub 2024 Aug 30. PMID 39213194

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 655 participants with hereditary amyloid transthyretin (hATTR) amyloidosis or wild-type ATTR (wtATTR) amyloidosis with cardiomyopathy took part in the study at 87 sites across 26 countries in North America, South America, Europe, Asia, and Australia. This study is still ongoing.
Pre-assignment Details: The study consists of 2 parts: Double-blind (DB) Period and Open-label Treatment Extension (OLE) Period. In the DB period, participants were randomized in a 1:1 ratio to receive vutrisiran or placebo and during the OLE Period, all participants receive vutrisiran. The DB period of the study has been completed while OLE period is still ongoing.
Groups:
- DB Period: Placebo: Participants in the DB period received vutrisiran matching placebo, subcutaneous (SC) injection, once every 3 months (q3M) for up to 36 months.
- DB Period: Vutrisiran: Participants in the DB period received vutrisiran, 25 mg, SC injection, q3M for up to 36 months.
- OLE Period: Placebo/Vutrisiran: Participants who received placebo in the DB period receive vutrisiran, 25 mg, SC injection, q3M for up to 24 months in the OLE period.
- OLE Period: Vutrisiran/Vutrisiran: Participants who received vutrisiran 25 mg in the DB period continue receiving vutrisiran, 25 mg, SC injection, q3M for up to 24 months in the OLE period.
Period: Double Blind Period
Arm/Group | DB Period: Placebo | DB Period: Vutrisiran | OLE Period: Placebo/Vutrisiran | OLE Period: Vutrisiran/Vutrisiran
Started | 329 | 326 | 0 | 0
Completed | 235 | 257 | 0 | 0
Not Completed | 94 | 69 | 0 | 0
Not completed — Death | 63 | 49 | 0 | 0
Not completed — Withdrawal by Subject | 16 | 11 | 0 | 0
Not completed — Adverse Event | 6 | 2 | 0 | 0
Not completed — Lost to Follow-up | 2 | 1 | 0 | 0
Not completed — Withdrawal by guardian | 0 | 2 | 0 | 0
Not completed — Reason Not Specified | 5 | 4 | 0 | 0
Not completed — Physician Decision | 2 | 0 | 0 | 0
Period: Open Label Extension Period
Arm/Group | DB Period: Placebo | DB Period: Vutrisiran | OLE Period: Placebo/Vutrisiran | OLE Period: Vutrisiran/Vutrisiran
Started | 0 | 0 | 221 | 241
Completed | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 221 | 241
Not completed — Death | 0 | 0 | 7 | 3
Not completed — Withdrawal by guardian | 0 | 0 | 1 | 0
Not completed — Participant Withdrew from Treatment but Ongoing in Safety Follow-up | 0 | 0 | 0 | 1
Not completed — Study Treatment Ongoing | 0 | 0 | 213 | 237

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) included all participants who were randomized and received any amount of study drug (vutrisiran or placebo). 1 participant randomized to placebo was not dosed and hence was excluded from FAS.
Groups:
- DB Period: Placebo: Participants in the DB period received vutrisiran matching placebo, SC injection, q3M for up to 36 months.
- Total: Total of all reporting groups
Arm/Group | DB Period: Placebo | DB Period: Vutrisiran | Total
Number analyzed (Participants) | 328 | 326 | 654
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.2 (6.3) | 75.5 (7.2) | 75.4 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 27 | 49
  Male | 306 | 299 | 605
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 22 | 38
  Not Hispanic or Latino | 304 | 298 | 602
  Unknown or Not Reported | 8 | 6 | 14
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 19 | 18 | 37
  Black or African American | 24 | 23 | 47
  White | 275 | 277 | 552
  Not reported | 8 | 6 | 14
  Other | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Composite Endpoint of All-Cause Mortality and Recurrent Cardiovascular (CV) Events (CV Hospitalizations and Urgent Heart Failure [HF] Visits) in the Overall Population
Description: All-cause mortality and recurrent CV events (CV hospitalizations and urgent HF visits) were compared between treatment groups using a modified Andersen-Gill model with a robust variance. All-cause mortality included heart transplantation and LVAD placement events along with deaths; recurrent CV events included CV hospitalizations and urgent HF visits. The number of participants with at least one CV event or all-cause mortality event have been reported here. No imputation was done for participants who dropped out early for the primary analysis of this composite outcome endpoint.
Time Frame: Up to Month 36
Population: FAS included all participants who were randomized and received any amount of study drug (vutrisiran or placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | DB Period: Placebo | DB Period: Vutrisiran
Number analyzed (Participants) | 328 | 326
Participants | 159 | 125
Statistical Analysis 1: Comparison: DB Period: Placebo vs DB Period: Vutrisiran; Analysis done using a modified Andersen-Gill model with a robust variance. The model included treatment group, ATTR amyloidosis disease type, New York Heart Association (NYHA) class, age group, and log-transformed baseline N-terminal pro-B-type natriuretic peptide (NT-proBNP) as covariates; Test type: Superiority; p = 0.0118, Modified Andersen-Gill Model; Hazard Ratio (HR) = 0.718, 95% CI 2-sided [0.555 to 0.929]

2. Primary Outcome: Composite Endpoint of All-Cause Mortality and Recurrent CV Events (CV Hospitalizations and Urgent HF Visits) in the Vutrisiran Monotherapy Subgroup
Description: as for outcome 1
Time Frame: Up to Month 36
Population: Vutrisiran Monotherapy Subgroup FAS included all participants who were not on tafamidis at the study baseline in the FAS. FAS included all participants who were randomized and received any amount of study drug (vutrisiran or placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | DB Period: Placebo | DB Period: Vutrisiran
Number analyzed (Participants) | 199 | 196
Participants | 105 | 76
Statistical Analysis 1: Comparison: DB Period: Placebo vs DB Period: Vutrisiran; Analysis done using a modified Andersen-Gill model with a robust variance. The model included treatment group, ATTR amyloidosis disease type, NYHA class, age group, and log-transformed baseline NT-proBNP as covariates; Test type: Superiority; p = 0.0162, Modified Andersen-Gill Model; Hazard Ratio (HR) = 0.672, 95% CI 2-sided [0.487 to 0.929]

3. Secondary Outcome: Change From Baseline in 6-Minute Walk Test (6-MWT) in the Overall Population
Description: The 6-MWT is an assessment of functional exercise capacity. Participants are instructed to walk back and forth along a flat, straight path, typically 30 meters in length, for a duration of 6 minutes. The total distance covered in meters is recorded at the end of 6 minutes. A longer distance reflects a better outcome. Analysis was based on the mixed-effect model of repeated measures (MMRM). Missing change values due to amyloidosis disease progression and death were imputed using sampling with replacement from the worst 10% of observed values, as specified in the statistical analysis plan (SAP).
Time Frame: Baseline to Month 30
Population: FAS included all participants who were randomized and received any amount of study drug (vutrisiran or placebo). Overall number analyzed is the number of participants with data available for analysis.
Measure: Least Squares Mean (Standard Error); unit: meters
Arm/Group | DB Period: Placebo | DB Period: Vutrisiran
Number analyzed (Participants) | 328 | 325
meters | -71.88 (4.79) | -45.42 (4.62)
Statistical Analysis 1: Comparison: DB Period: Placebo vs DB Period: Vutrisiran; Analysis done using MMRM with baseline 6-MWT as a covariate and fixed effect terms including treatment group, visit, treatment-by-visit interaction, baseline tafamidis use, treatment-by-baseline tafamidis use interaction, type of ATTR amyloidosis, and age group. Missing change values due to amyloidosis disease progression and death were imputed using sampling with replacement from the worst 10% of observed values, as specified in the SAP; Test type: Superiority; p = 0.0000797, MMRM; Least Square (LS) Mean Difference = 26.46, 95% CI 2-sided [13.38 to 39.55], Standard Error of Mean 6.66

4. Secondary Outcome: Change From Baseline in 6-MWT in the Vutrisiran Monotherapy Subgroup
Description: The 6-MWT is an assessment of functional exercise capacity. Participants are instructed to walk back and forth along a flat, straight path, typically 30 meters in length, for a duration of 6 minutes. The total distance covered in meters is recorded at the end of 6 minutes. A longer distance reflects a better outcome. Analysis was based on the MMRM. Missing change values due to amyloidosis disease progression and death were imputed using sampling with replacement from the worst 10% of observed values, as specified in the SAP.
Time Frame: Baseline to Month 30
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: meters
Arm/Group | DB Period: Placebo | DB Period: Vutrisiran
Number analyzed (Participants) | 199 | 196
meters | -91.78 (6.39) | -59.69 (6.60)
Statistical Analysis 1: Comparison: DB Period: Placebo vs DB Period: Vutrisiran; Analysis done using MMRM with baseline 6-MWT as a covariate and fixed effect terms including treatment group, visit, treatment-by-visit interaction, type of ATTR amyloidosis, and age group. Missing change values due to amyloidosis disease progression and death were imputed using sampling with replacement from the worst 10% of observed values, as specified in the SAP; Test type: Superiority; p = 0.0005, MMRM; LS Mean Difference = 32.09, 95% CI 2-sided [14.03 to 50.15], Standard Error of Mean 9.19

5. Secondary Outcome: Change From Baseline in the Kansas City Cardiomyopathy Questionnaire Overall Summary (KCCQ-OS) Score in the Overall Population
Description: The KCCQ is a 23-item self-administered questionnaire quantifying 6 domains (symptoms [frequency and burden], physical function, quality of life (QoL), social limitation, self-efficacy, and symptom stability) and 2 summary scores (clinical and overall summary [OS]). Scores were generated for each domain and transformed to a range of 0-100, in which higher scores reflect better health status. KCCQ- overall summary score was average of domains- physical function, total symptoms (average of symptom frequency and burden), QoL, and social limitation, and transformed to a single score which ranged from 0 (worst) - 100 (the best possible status), where the higher score reflected better health status. Analysis was based on the MMRM.
Time Frame: Baseline to Month 30
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | DB Period: Placebo | DB Period: Vutrisiran
Number analyzed (Participants) | 327 | 325
score on a scale | -15.49 (1.26) | -9.68 (1.19)
Statistical Analysis 1: Comparison: DB Period: Placebo vs DB Period: Vutrisiran; Analysis done using MMRM with baseline KCCQ-OS as a covariate and fixed effect terms including treatment group, visit, treatment-by-visit interaction, baseline tafamidis use, treatment-by-baseline tafamidis use interaction, type of ATTR amyloidosis, and age group. Missing change values due to death were imputed using sampling with replacement from the worst 10% of observed values, as specified in the SAP; Test type: Superiority; p = 0.0008, MMRM; LS Mean Difference = 5.8, 95% CI 2-sided [2.40 to 9.20], Standard Error of Mean 1.73

6. Secondary Outcome: Change From Baseline in the KCCQ-OS Score in the Vutrisiran Monotherapy Subgroup
Description: The KCCQ is a 23-item self-administered questionnaire quantifying 6 domains (symptoms [frequency and burden], physical function, QoL, social limitation, self-efficacy, and symptom stability) and 2 summary scores (clinical and OS). Scores were generated for each domain and transformed to a range of 0-100, in which higher scores reflect better health status. KCCQ- overall summary score was average of domains- physical function, total symptoms (average of symptom frequency and burden), QoL, and social limitation, and transformed to a single score which ranged from 0 (worst) - 100 (the best possible status), where the higher score reflected better health status. Analysis was based on the MMRM.
Time Frame: Baseline to Month 30
Population: Vutrisiran Monotherapy Subgroup FAS included all participants who were not on tafamidis at the study baseline in the FAS. Overall number analyzed is the number of participants with data available for analysis.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | DB Period: Placebo | DB Period: Vutrisiran
Number analyzed (Participants) | 198 | 195
score on a scale | -19.47 (1.73) | -10.78 (1.66)
Statistical Analysis 1: Comparison: DB Period: Placebo vs DB Period: Vutrisiran; Analysis done using MMRM with baseline KCCQ-OS as a covariate and fixed effect terms including treatment group, visit, treatment-by-visit interaction, type of ATTR amyloidosis, and age group. Missing change values due to death were imputed using sampling with replacement from the worst 10% of observed values, as specified in the SAP; Test type: Superiority; p = 0.0003, MMRM; LS Mean Difference = 8.69, 95% CI 2-sided [3.98 to 13.40], Standard Error of Mean 2.4

7. Secondary Outcome: All-cause Mortality in the Overall Population and Vutrisiran Monotherapy Subgroup
Description: All-cause mortality also included heart transplantation and LVAD placement events along with deaths; recurrent CV events included CV hospitalizations and urgent HF visits.
Time Frame: Up to 42 months
Reporting Status: Not Posted, anticipated posting 2027-12

8. Secondary Outcome: Percentage of Participants With Change in NYHA Class at Month 30 in the Overall Population
Description: NYHA class is a clinical assessment of symptoms resulting from heart failure. In NYHA functional classification system places participants in 1 of 4 categories based on limitations of physical activity. Class I denotes no symptoms and no limitation of physical activity; II, slight limitation, resulting in symptoms with ordinary physical activity; III, marked limitation, resulting in symptoms with less than ordinary physical activity; and IV, symptoms at rest. Here, the participants with a change in NYHA class have been reported in two categories:
  1) participants who had no change or had improvement in the NYHA class (lower class) from baseline and 2) participants who had a worsened NYHA class from baseline (higher class).
  Values have been rounded off to a single decimal.
Time Frame: Baseline to Month 30
Population: FAS included all participants who were randomized and received any amount of study drug (vutrisiran or placebo).
Measure: Number; unit: percentage of participants
Arm/Group | DB Period: Placebo | DB Period: Vutrisiran
Number analyzed (Participants) | 328 | 326
percentage of participants
  Stable or improved from baseline | 60.5 | 67.8
  Worsened from baseline | 39.5 | 32.2
Statistical Analysis 1: Comparison: DB Period: Placebo vs DB Period: Vutrisiran; Test type: Superiority; p = 0.0217, Cochran-Mantel-Haenszel; Missing change value in NYHA Class due to death were imputed as worsened. All other missing were imputed using multiple imputation approach; Mean Difference = 8.7, 95% CI 2-sided [1.3 to 16.1] — Adjusted difference in percentage of stable or improved (vutrisiran - placebo) participants was estimated. Adjusted difference, 95% CI, and p-value were derived from multiple imputation procedure by combining estimates per Rubin's rules

9. Secondary Outcome: Percentage of Participants With Change in NYHA Class at Month 30 in the Vutrisiran Monotherapy Subgroup
Description: as for outcome 8
Time Frame: Baseline to Month 30
Population: Vutrisiran Monotherapy Subgroup FAS included all participants who were not on tafamidis at the study baseline in the FAS.
Measure: Number; unit: percentage of participants
Arm/Group | DB Period: Placebo | DB Period: Vutrisiran
Number analyzed (Participants) | 199 | 196
percentage of participants
  Stable or improved from baseline | 56.4 | 66.3
  Worsened from baseline | 43.6 | 33.7
Statistical Analysis 1: Comparison: DB Period: Placebo vs DB Period: Vutrisiran; Test type: Superiority; p = 0.0121, Cochran-Mantel-Haenszel; [statistical method as in outcome 8, analysis 1]; Mean Difference = 12.5, 95% CI 2-sided [2.7 to 22.2] — [estimate comment as in outcome 8, analysis 1]

ADVERSE EVENTS:
Time Frame: Up to Month 36
Description: Safety Analysis Set included all participants who received any amount of study drug. 1 participant randomized to placebo was not dosed and not included in the analysis. DB period is completed and data collected during the DB period are reported here. Data collection for the OLE period is still ongoing. Adverse event data for the OLE period will be reported one year after the study completion date.
Arm/Group | DB Period: Placebo | DB Period: Vutrisiran
All-Cause Mortality (participants affected / at risk) | 63/328 | 49/326
Serious Adverse Events (participants affected / at risk) | 220/328 | 201/326
Other Adverse Events (participants affected / at risk) | 303/328 | 293/326
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DB Period: Placebo (N=328) | DB Period: Vutrisiran (N=326)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Blood loss anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hilar lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymphadenopathy mediastinal (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Nephrogenic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 2 (2) | 3 (3)
Acute left ventricular failure (Cardiac disorders) | 1 (1) | 2 (2)
Acute myocardial infarction (Cardiac disorders) | 3 (3) | 4 (5)
Angina pectoris (Cardiac disorders) | 2 (2) | 0 (0)
Angina unstable (Cardiac disorders) | 1 (1) | 1 (1)
Aortic valve stenosis (Cardiac disorders) | 0 (0) | 1 (1)
Arrhythmia (Cardiac disorders) | 3 (3) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 20 (27) | 26 (29)
Atrial flutter (Cardiac disorders) | 9 (9) | 9 (10)
Atrial tachycardia (Cardiac disorders) | 3 (8) | 1 (1)
Atrial thrombosis (Cardiac disorders) | 1 (1) | 0 (0)
Atrioventricular block (Cardiac disorders) | 3 (3) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 5 (5) | 6 (6)
Atrioventricular block first degree (Cardiac disorders) | 0 (0) | 3 (3)
Atrioventricular block second degree (Cardiac disorders) | 1 (1) | 1 (1)
Bifascicular block (Cardiac disorders) | 1 (1) | 1 (1)
Bradycardia (Cardiac disorders) | 7 (8) | 3 (3)
Bundle branch block left (Cardiac disorders) | 0 (0) | 1 (1)
Bundle branch block right (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac amyloidosis (Cardiac disorders) | 3 (4) | 1 (1)
Cardiac arrest (Cardiac disorders) | 2 (2) | 2 (2)
Cardiac failure (Cardiac disorders) | 57 (94) | 38 (70)
Cardiac failure acute (Cardiac disorders) | 18 (21) | 13 (16)
Cardiac failure chronic (Cardiac disorders) | 4 (4) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 15 (21) | 4 (4)
Cardiac perforation (Cardiac disorders) | 0 (0) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 7 (8) | 4 (4)
Cardiorenal syndrome (Cardiac disorders) | 0 (0) | 2 (2)
Chronotropic incompetence (Cardiac disorders) | 1 (1) | 0 (0)
Conduction disorder (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 4 (4) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 1 (1)
Hypertensive heart disease (Cardiac disorders) | 0 (0) | 1 (1)
Left ventricular dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Left ventricular failure (Cardiac disorders) | 1 (1) | 2 (2)
Low cardiac output syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Microvascular coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 0 (0) | 2 (2)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 2 (2) | 0 (0)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Sinus node dysfunction (Cardiac disorders) | 1 (1) | 2 (2)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Tricuspid valve incompetence (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 1 (1) | 2 (2)
Ventricular fibrillation (Cardiac disorders) | 2 (2) | 1 (1)
Ventricular tachyarrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 8 (9) | 8 (9)
Cystic fibrosis (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Deafness neurosensory (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 (0) | 1 (1)
Thyroid mass (Endocrine disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 1 (2) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 1 (1)
Visual impairment (Eye disorders) | 0 (0) | 1 (1)
Abdominal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Barrett's oesophagus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 2 (2) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 4 (4) | 1 (1)
Gastrointestinal vascular malformation haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Incarcerated inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 1 (1)
Intra-abdominal fluid collection (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 2 (2) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Obstructive pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal food impaction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ulcerative gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 2 (2) | 1 (1)
Cardiac death (General disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 7 (8) | 4 (5)
Complication associated with device (General disorders) | 0 (0) | 1 (1)
Death (General disorders) | 3 (3) | 0 (0)
Disease progression (General disorders) | 5 (5) | 0 (0)
Drowning (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 2 (2) | 1 (1)
General physical health deterioration (General disorders) | 1 (2) | 0 (0)
Generalised oedema (General disorders) | 1 (1) | 0 (0)
Hernia pain (General disorders) | 2 (2) | 0 (0)
Implant site haematoma (General disorders) | 0 (0) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 2 (2) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 2 (2)
Oedema (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Organ failure (General disorders) | 0 (0) | 1 (1)
Peripheral swelling (General disorders) | 1 (1) | 0 (0)
Physical deconditioning (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 2 (2)
Cholecystitis acute (Hepatobiliary disorders) | 2 (2) | 1 (1)
Cholecystitis chronic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (3) | 1 (2)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0)
Ischaemic hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Anti-neutrophil cytoplasmic antibody positive vasculitis (Immune system disorders) | 1 (1) | 0 (0)
Adenovirus infection (Infections and infestations) | 0 (0) | 1 (1)
Appendicitis perforated (Infections and infestations) | 0 (0) | 1 (1)
Arthritis bacterial (Infections and infestations) | 1 (1) | 1 (1)
Bacteraemia (Infections and infestations) | 3 (3) | 0 (0)
Bacterial infection (Infections and infestations) | 2 (2) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Bursitis infective (Infections and infestations) | 0 (0) | 2 (2)
COVID-19 (Infections and infestations) | 5 (5) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 2 (2) | 1 (1)
Cellulitis (Infections and infestations) | 4 (4) | 4 (4)
Cerebral malaria (Infections and infestations) | 0 (0) | 1 (1)
Chronic sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 2 (2) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 1 (1)
Cystitis escherichia (Infections and infestations) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 2 (3) | 1 (1)
Diverticulitis (Infections and infestations) | 4 (5) | 0 (0)
Emphysematous cholecystitis (Infections and infestations) | 1 (3) | 0 (0)
Enterococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Gallbladder abscess (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis norovirus (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0)
Implant site infection (Infections and infestations) | 0 (0) | 1 (1)
Infectious pleural effusion (Infections and infestations) | 1 (1) | 0 (0)
Infective corneal ulcer (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Medical device site infection (Infections and infestations) | 1 (1) | 0 (0)
Meningitis (Infections and infestations) | 0 (0) | 1 (1)
Ophthalmic herpes simplex (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 10 (11) | 12 (13)
Post procedural infection (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 3 (3) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0)
Respiratory syncytial virus bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 2 (2) | 1 (2)
Sepsis (Infections and infestations) | 3 (3) | 6 (6)
Septic phlebitis (Infections and infestations) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 3 (3) | 3 (3)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Soft tissue infection (Infections and infestations) | 1 (1) | 0 (0)
Spinal cord infection (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal sepsis (Infections and infestations) | 1 (1) | 2 (2)
Tracheobronchitis (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 4 (4) | 2 (2)
Urosepsis (Infections and infestations) | 0 (0) | 6 (6)
Acetabulum fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Carbon monoxide poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Complications of transplanted heart (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 8 (8) | 6 (6)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Flatback syndrome (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fractured coccyx (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 4 (4)
Intentional overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Multiple injuries (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Post procedural bile leak (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Respiratory fume inhalation disorder (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (2)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Seroma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (2) | 1 (1)
Spinal cord injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Sternal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ulnar nerve injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Urinary retention postoperative (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Cardiovascular evaluation (Investigations) | 1 (1) | 0 (0)
Catheterisation cardiac (Investigations) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Fluid retention (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypervolaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 7 (7) | 3 (3)
Hypovolaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Metabolic alkalosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Haematoma muscle (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Mobility decreased (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 8 (10) | 10 (10)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (2)
Abdominal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Angiosarcoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (5) | 1 (4)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lentigo maligna (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Malignant melanoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Rhabdomyosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Spinal meningioma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Spindle cell sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Squamous cell carcinoma of head and neck (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Altered state of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0)
Brain injury (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral arteriosclerosis (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral artery embolism (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 1 (1)
Cerebral infarction (Nervous system disorders) | 3 (3) | 2 (2)
Cerebral ischaemia (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrospinal fluid leakage (Nervous system disorders) | 0 (0) | 1 (2)
Cerebrovascular accident (Nervous system disorders) | 4 (4) | 2 (2)
Cerebrovascular disorder (Nervous system disorders) | 0 (0) | 1 (1)
Cubital tunnel syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Dementia (Nervous system disorders) | 0 (0) | 1 (1)
Dementia Alzheimer's type (Nervous system disorders) | 1 (1) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Embolic stroke (Nervous system disorders) | 1 (1) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Hemiparesis (Nervous system disorders) | 0 (0) | 1 (1)
Hepatic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 3 (3) | 1 (1)
Metabolic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Motor neurone disease (Nervous system disorders) | 0 (0) | 1 (2)
Nerve compression (Nervous system disorders) | 0 (0) | 1 (1)
Parkinson's disease (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 2 (2) | 1 (1)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 1 (1) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 7 (8) | 8 (10)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Uraemic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Vertebrobasilar stroke (Nervous system disorders) | 0 (0) | 1 (1)
Device dislocation (Product Issues) | 0 (0) | 1 (1)
Device malfunction (Product Issues) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 1 (1)
Hallucinations, mixed (Psychiatric disorders) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 10 (13) | 11 (12)
Bladder stenosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 2 (2) | 1 (1)
Cystitis haemorrhagic (Renal and urinary disorders) | 1 (1) | 0 (0)
Diabetic nephropathy (Renal and urinary disorders) | 0 (0) | 1 (1)
End stage renal disease (Renal and urinary disorders) | 0 (0) | 2 (2)
Haematuria (Renal and urinary disorders) | 1 (1) | 4 (5)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal impairment (Renal and urinary disorders) | 2 (2) | 0 (0)
Renal tubular dysfunction (Renal and urinary disorders) | 0 (0) | 1 (1)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Urethral perforation (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 5 (6) | 3 (3)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 2 (2)
Peyronie's disease (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Prostatic obstruction (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pharyngeal haematoma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 5 (8)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Loss of personal independence in daily activities (Social circumstances) | 1 (1) | 0 (0)
Cardiac pacemaker insertion (Surgical and medical procedures) | 0 (0) | 3 (3)
Cardioversion (Surgical and medical procedures) | 1 (1) | 0 (0)
Coronary angioplasty (Surgical and medical procedures) | 0 (0) | 1 (1)
Diverticulectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Hip arthroplasty (Surgical and medical procedures) | 0 (0) | 1 (1)
Implantable defibrillator replacement (Surgical and medical procedures) | 0 (0) | 1 (1)
Lymphadenectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Transcatheter aortic valve implantation (Surgical and medical procedures) | 0 (0) | 1 (1)
Wound treatment (Surgical and medical procedures) | 1 (1) | 0 (0)
Aortic dilatation (Vascular disorders) | 0 (0) | 1 (1)
Aortic dissection (Vascular disorders) | 0 (0) | 1 (1)
Aortic stenosis (Vascular disorders) | 1 (1) | 0 (0)
Atheroembolism (Vascular disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 1 (2)
Dry gangrene (Vascular disorders) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 2 (2)
Hypotension (Vascular disorders) | 3 (3) | 5 (5)
Orthostatic hypotension (Vascular disorders) | 2 (2) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 2 (2) | 0 (0)
Peripheral artery occlusion (Vascular disorders) | 1 (1) | 0 (0)
Shock haemorrhagic (Vascular disorders) | 0 (0) | 1 (1)
Subclavian vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DB Period: Placebo (N=328) | DB Period: Vutrisiran (N=326)
Anaemia (Blood and lymphatic system disorders) | 16 (16) | 19 (20)
Atrial fibrillation (Cardiac disorders) | 58 (65) | 59 (78)
Atrial flutter (Cardiac disorders) | 17 (21) | 24 (26)
Cardiac failure (Cardiac disorders) | 105 (161) | 79 (103)
Cardiac failure congestive (Cardiac disorders) | 17 (18) | 8 (9)
Palpitations (Cardiac disorders) | 18 (18) | 4 (4)
Hypothyroidism (Endocrine disorders) | 17 (17) | 11 (11)
Constipation (Gastrointestinal disorders) | 42 (53) | 33 (35)
Diarrhoea (Gastrointestinal disorders) | 30 (34) | 15 (16)
Nausea (Gastrointestinal disorders) | 26 (28) | 9 (10)
Chest pain (General disorders) | 23 (29) | 17 (20)
Fatigue (General disorders) | 43 (56) | 27 (32)
Oedema peripheral (General disorders) | 25 (28) | 33 (40)
COVID-19 (Infections and infestations) | 97 (104) | 86 (92)
Cellulitis (Infections and infestations) | 19 (21) | 16 (18)
Pneumonia (Infections and infestations) | 17 (17) | 15 (17)
Upper respiratory tract infection (Infections and infestations) | 24 (27) | 16 (17)
Urinary tract infection (Infections and infestations) | 36 (45) | 32 (44)
Fall (Injury, poisoning and procedural complications) | 66 (103) | 39 (58)
Skin laceration (Injury, poisoning and procedural complications) | 18 (22) | 13 (14)
Gout (Metabolism and nutrition disorders) | 51 (77) | 47 (78)
Hypervolaemia (Metabolism and nutrition disorders) | 21 (36) | 15 (16)
Hypokalaemia (Metabolism and nutrition disorders) | 25 (33) | 16 (18)
Arthralgia (Musculoskeletal and connective tissue disorders) | 38 (45) | 33 (49)
Back pain (Musculoskeletal and connective tissue disorders) | 31 (37) | 36 (41)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 24 (28) | 20 (23)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 19 (24) | 14 (15)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 14 (16) | 21 (22)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 32 (48) | 27 (40)
Carpal tunnel syndrome (Nervous system disorders) | 19 (20) | 10 (11)
Dizziness (Nervous system disorders) | 43 (52) | 32 (36)
Headache (Nervous system disorders) | 20 (22) | 9 (12)
Paraesthesia (Nervous system disorders) | 18 (22) | 8 (8)
Syncope (Nervous system disorders) | 23 (29) | 14 (14)
Insomnia (Psychiatric disorders) | 22 (23) | 18 (18)
Acute kidney injury (Renal and urinary disorders) | 19 (23) | 22 (25)
Chronic kidney disease (Renal and urinary disorders) | 17 (20) | 16 (17)
Haematuria (Renal and urinary disorders) | 26 (33) | 20 (22)
Cough (Respiratory, thoracic and mediastinal disorders) | 27 (28) | 24 (26)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 48 (61) | 42 (47)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 20 (22) | 15 (17)
Pruritus (Skin and subcutaneous tissue disorders) | 21 (24) | 13 (13)
Hypotension (Vascular disorders) | 22 (23) | 8 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2024-02-12): https://cdn.clinicaltrials.gov/large-docs/49/NCT04153149/Prot_002.pdf
  • Statistical Analysis Plan (2024-05-30): https://cdn.clinicaltrials.gov/large-docs/49/NCT04153149/SAP_003.pdf